CLINICAL TRIAL: NCT06054750
Title: Testing Regional anesthesia Techniques For Up And Early Discharge Following Knee arthroplasty: Quality Of Recovery Through Patient Reporting - a Feasibility Study
Brief Title: Testing Regional anesthesia Techniques For Up And Early Discharge Following Knee arthroplasty - a Feasibility Study
Acronym: TRUE KnORTH 2
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRUE KnORTH 2.0
Record Dates: First submitted 2023-09-11; First posted 2023-09-26 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-09

CONDITIONS: Arthroplasty, Replacement, Knee
MeSH Terms: interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pharmacy will have access to the randomization scheme. All other members of the study team are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cACB active (Experimental): Periarticular joint injection (medication) + single shot adductor canal block (medication) + adductor canal catheter infusion (medication)
  Interventions: Drug: Ropivacaine
- cACB sham (Placebo Comparator): Periarticular joint injection (medication) + single shot adductor canal block (medication) + adductor canal catheter infusion (normal saline)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ropivacaine — 800 mg ropivacaine in continuous infusion adductor canal block (400 mL total volume)
  Arms: cACB active
Drug: Normal saline — 400 mL normal saline in continuous infusion adductor canal block (400 mL total volume)
  Arms: cACB sham

SUMMARY:
To assess feasibility of a a trial investigation postoperative patient-reported quality of recovery after total knee arthroplasty (TKA) with periarticular joint injection (PAI) ± single shot adductor canal block with or without adductor canal catheter infusion.

DETAILED DESCRIPTION:
Knee osteoarthritis (KOA) is a leading cause of chronic knee pain and disability, with a lifetime prevalence of 45%. Treatment for symptomatic KOA includes physical therapy, oral anti-inflammatory medications and intra-articular steroid injections, with total knee arthroplasty (TKA) (or knee replacement) as the definitive treatment. Acute postoperative pain is common after TKA, leading to increased opioid consumption and increased hospital length of stay. Pain control following TKA has been investigated with interventions such as intrathecal morphine, nerve blocks, and periarticular joint injection (PAI). PAI and adductor canal block are well-established techniques used both in combination or in isolation in the management of postoperative pain for patients undergoing TKA. The aim of this study is to assess postoperative patient-reported quality of recovery after TKA with PAI and single shot adductor canal block with or without adductor canal catheter infusion.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients presenting for a primary TKA.

Exclusion Criteria:

* Age <18 years;
* Body mass index ≥45 kg/m2;
* Weight <80 kg;
* Deemed unsuitable for regional anesthesia;
* Planned general anesthesia;
* Hepatic insufficiency/Intolerance to acetaminophen;
* Renal insufficiency (defined by estimated glomerular filtration rate <60 mL/min/1.73 m2);
* Chronic opioid use (individuals requiring the equivalent of 1 mg or more of intravenous morphine, or 3 mg or more of oral morphine per hour for greater than 1 month);
* Allergy or intolerance to study medications (listed under 'Spinal and Adductor Canal Block') or trial medications listed in "Postoperative" section and "standard prescription"
* Clinical Frailty Scale score ≥4;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery-15 Survey scores | Postoperative day 0 (2 hours postoperatively), and morning of postoperative days 1, 2 and 3
  Patient-reported Quality of Recovery scores, where higher scores indicate better quality of recovery

SECONDARY OUTCOMES:
Quality of Recovery-15 Survey scores | Postoperative days 10 and 42
  Patient-reported Quality of Recovery scores, where higher scores indicate better quality of recovery
Brief Pain Inventory - Pain Interference scores | Postoperative days 1, 2 and 3 in the morning
  On a scale of 0-10, where 0=Does not interfere and 10=Completely interferes, Patients will rate how much their pain interferes with: General activity, Mood, Walking ability, Normal work including housework, Relations with other people, Sleep, and Enjoyment of life
Pain Numerical Rating Scale at rest | Postoperative Day 0 (2 hours postoperatively), and morning of postoperative days 1, 2 and 3
  Patient-reported pain measured on an 11-point scale from 0 [no pain] to 10 [worst pain imaginable]
Pain Numerical Rating Scale with activity | Postoperative Day 0 (2 hours postoperatively), and morning of postoperative days 1, 2 and 3 after physiotherapy
  Patient-reported pain measured on an 11-point scale from 0 [no pain] to 10 [worst pain imaginable]
Functional Recovery: Range of motion | Postoperative Day 0 (2 hours postoperatively), and morning of postoperative days 1, 2 and 3 after physiotherapy
  Flexion and Extension range of motion measured in degrees
Functional Recovery: Time to reach discharge criteria | Postoperative Day 0 (2 hours postoperatively), and morning of postoperative days 1, 2 and 3 after physiotherapy
  Physiotherapist to assess when patient meets discharge criteria (measured in half days)
Functional Recovery: Timed Up and Go test | Postoperative day 42
  Time it takes for patient to stand up from sitting in a chair, walk 3 meters, then turn and walk back to chair and sit down, measured in seconds
Frequency of opioid-related side effects (vomiting and nausea) | Up to 3 days
  Number of vomiting events or complaints of nausea noted in nursing notes
Narcotic consumption in hospital | Up to 3 days
  total amount and route of administration collected from routine and PRN opioid use in PACU and on surgical floor - measured in mg of oral morphine equivalence
Narcotic consumption at home | Postoperative day 42
  Post-discharge opioid consumption will be tracked with pill count on POD 1 or 2, 3 POD10 (± 2 days), and POD42 (± 2 days); on POD 42 - patient to show study nurse how many pills remain to ensure reporting accuracy
Complications | Postoperative days 10 and 42
  i. return to hospital once discharged for non-analgesic reasons ii. require more pain medications outside of prescription given

CONTACTS AND LOCATIONS:
Locations (1):
- St Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided